CLINICAL TRIAL: NCT00678431
Title: A Single Center, Multi-site, Randomized, Double-blind, Placebo-controlled Trial of Resveratrol With Glucose and Malate (RGM) to Slow the Progression of Alzheimer's Disease
Brief Title: Randomized Trial of a Nutritional Supplement in Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Alzheimer's Association (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0553-06-071
Record Dates: First submitted 2008-01-07; First posted 2008-05-15 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Dementia; Nutritional Supplement; Resveratrol
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Resveratrol; Glucose; malic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Placebo Comparator): Liquid placebo
  Interventions: Dietary Supplement: Placebo
- Arm 2 (Experimental): Liquid Resveratrol with Glucose, and Malate
  Interventions: Dietary Supplement: Resveratrol with Glucose, and Malate

INTERVENTIONS:
Dietary Supplement: Resveratrol with Glucose, and Malate — Dietary supplement delivered in grape juice
  Arms: Arm 2
Dietary Supplement: Placebo — Liquid placebo
  Arms: Arm 1

SUMMARY:
Alzheimer's disease (AD), one of the leading causes of morbidity and mortality in the elderly is characterized by progressive cognitive decline and certain neuropathological features.

Currently, there is great interest in the well-documented mitochondrial (oxidative) lesion in AD. Disturbed oxidative metabolism is a well described abnormality in AD. Several observational studies have shown that moderate consumption of wine is associated with a lower incidence of Alzheimer's disease (Truelsen et al., 2002; Luchsinger et al., 2004). Wine is enriched in antioxidant compounds with potential neuroprotective activities. In the early 1990s the presence of Resveratrol in red wine was detected where it is suspected to afford antioxidant and neuroprotective properties (Miller and Rice-Evans, 1995).

Blass and Gordon (2004) have demonstrated positive effects in AD with an oral preparation of glucose, malate and resveratrol. Glucose is the physiological precursor of the substrates of oxidative metabolism in the brain, malate is a primer of the energy-providing Krebs-cycle. Glucose and malate therefore can provide reducing equivalents (electrons) to regenerate the reduced form of resveratrol, and do so under the normal regulation of brain cell metabolism. All three ingredients are classified by the FDA as Generally Recognized As Safe.

DETAILED DESCRIPTION:
Subjects will be assessed by their capacity to consent by a psychiatrist independent of this study. Subjects who are determined to have capacity will sign consent. For subjects determined to lack capacity consent will be obtained from their surrogate. Subjects lacking in capacity must nonetheless provide verbal assent to participation in this study. After informed consent is obtained, subjects will be screened for eligibility to participate in the study. Screening comprises of medical history, physical exam, neurological exam, and a MMSE.

All of the above are performed for research purposes. Further evaluation of medical problems that are identified in the course of screening will be obtained as part of standard clinical care. For example, if an abnormality requiring further evaluation is detected on blood tests the subsequent evaluation will be conducted as standard clinical care.

Subjects who meet eligibility criteria will be baseline within 4 weeks. Eligible subjects will not be asked to stop any medication they may currently be on before the study begins. Eligible subjects will be randomized to receive either a mixture of glucose, malate and resveratrol (RGM) or placebo. At baseline, medical history, physical exam, cognitive tests are obtained. An ECG and a panel consisting CBC, electrolytes, liver and renal function tests will be drawn at the screening visit. Clinical information is obtained from the identified caregiver. The study drug (RGM or placebo, depending on which group the subject is randomly assigned to) is dispensed at baseline. Follow up visits at months 3, 6, 9, and 12 months require physical exam and some cognitive measures. At Month 12 a neurological exam will be performed. Adverse events are collected at each visit. Medication compliance is assessed at months 3, 6, 9, and 12 months and unused study drug is retrieved. At Month 12 unused study drug is retrieved and no more study drug is dispensed. Clinical information is obtained from the caregiver at each visit. At the Month 12 visit, a questionnaire will be completed by the study staff, subject and study partner to assess the adequacy of medication blinding. As noted all of the above tests and procedures are part of the research protocol. At study termination the subject will be referred to ongoing clinical care as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Consenting individuals as defined by IRB guidelines
2. NINCDS/ADRDA criteria for probable AD
3. Community dwelling
4. Age: greater than or equal to 50 years
5. MMSE between 12 and 26, inclusive
6. Stable medical condition for 3 months prior to screening visit
7. Stable doses of (non excluded) medications with central nervous system activity for 4 weeks prior to the screening visit (For cholinesterase inhibitors there should be no plan of dose escalation)
8. Physically acceptable for this study as confirmed by medical history, physical exam, neurologic exam and clinical laboratory tests
9. Supervision available for administration of study medications
10. Study partner to accompany subject to all scheduled visits and complete informant-based assessments.
11. Fluent in English or Spanish
12. Modified Hachinski < 4
13. CT or MRI since onset of memory impairment demonstrating absence of clinically significant focal lesion (One lacune in a non-critical brain region is acceptable)
14. Able to complete baseline assessments
15. 6 years of education, or work history sufficient to exclude mental retardation
16. Able to ingest oral medication

Exclusion Criteria:

1. Active liver disease or persistent elevation in serum transaminase
2. Severe renal disease
3. - Hx of diabetes mellitus (both insulin-dependent and non-insulin-dependent) or blood glucose >150 mg/dl
4. Active neoplastic disease (skin tumors other than melanoma are not exclusionary; subjects with stable prostate cancer or other stable cancers may be included at the discretion of the PI (Sano))
5. Use of another investigational agent within 2 months of the screening visit
6. History of clinically significant stroke
7. Current evidence or history in the past 2 years of seizures, head injury with loss of consciousness and/or immediate confusion after the injury
8. Current DSM-IV criteria-based diagnosis for major psychiatric disorder including psychosis, major depression, bipolar disorder, alcohol or substance abuse.
9. Blindness, deafness, language difficulties or any other disability which may interfere with testing ability
10. In female subjects, no history of menopause
11. Use of medications containing aluminum hydroxide, including anti-ulcer antacids such as Alternagel, Amphojel, Alu-tab, Maalox and Mylanta

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Alzheimer Disease Assessment Scale (ADAScog) | one year

SECONDARY OUTCOMES:
CGIC | one year

CONTACTS AND LOCATIONS:
Overall Officials: Mary Sano, PhD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

REFERENCES:
- [Derived] Zhu CW, Grossman H, Neugroschl J, Parker S, Burden A, Luo X, Sano M. A randomized, double-blind, placebo-controlled trial of resveratrol with glucose and malate (RGM) to slow the progression of Alzheimer's disease: A pilot study. Alzheimers Dement (N Y). 2018 Nov 9;4:609-616. doi: 10.1016/j.trci.2018.09.009. eCollection 2018. PMID 30480082